CLINICAL TRIAL: NCT06295887
Title: Development, Application, and Educational Efficacy of Medical Education Program Using Virtual Reality Technology
Brief Title: Educational Efficacy of VR vs. Simulator in Emergency Medical Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Sun Jung Myung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-2402
Record Dates: First submitted 2024-02-13; First posted 2024-03-06 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Simulation Training
Keywords: Emergency care performance

STUDY DESIGN:
Intervention Model Description: control group vs. test group, 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The test group wears an HMD (head-mounted display) and participates in a simulation program using VR. They experience both easy and difficult cases using VR. After the simulation session, a debriefing session will be provided.
  Interventions: Other: Educational Program using VR or simulator designed to improve medical intern's performance managing emergency situation
- Control group (Active Comparator): The control group participates in simulation training using Sim-man, and the scenarios are the same in both the control and the test groups (easy cases and difficult cases).
  After the simulation session, a debriefing session will be provided.
  Interventions: Other: Educational Program using VR or simulator designed to improve medical intern's performance managing emergency situation

INTERVENTIONS:
Other: Educational Program using VR or simulator designed to improve medical intern's performance managing emergency situation — Simulation program using VR or simulator that mimics patient's desaturation

SUMMARY:
It has not been revealed which is more effective: an education program using virtual reality technology or a simulation education program using Sim-man.

In this study, the participants are new doctors who graduated from medical school and started working as interns at hospitals. The participants were divided into two groups. One group received a training program using virtual reality technology, and the other group received simulation training using Sim-man. The investigators would like to compare the increase in confidence and satisfaction before and after training.

After the classes and surveys are completed for each group, the participants will be able to receive other educational methods if they wish.

DETAILED DESCRIPTION:
- The educational program was designed for participants to experience an emergency setting where a patient's oxygen saturation falls. The scenario starts with the decrease in the patient's oxygen saturation and the patient's condition could be changed according to the intern's management. The scenario includes various situations in which oxygen saturation could decrease, and the patient's condition changes depending on the expected responses of participants.

The scenario has been revised and supplemented through expert meetings.

* Experience two types of cases: an easy case where the patient's condition improves just by connecting an oxygen line, and a difficult case where the patient's condition does not improve even after connecting an oxygen line.
* A training program is prepared before the interns start work. The participants are divided into two groups (test group and control group). The test group wears an HMD (head-mounted display) and experiences both easy and difficult cases.
* The control group participates in simulation training using Sim-man, and the scenarios are the same for the test group (easy cases and difficult cases).
* Training on coping skills is provided through debriefing after VR and simulation.
* After completing the assigned program, participants can take the program that was not assigned to them if they wish.
* Both the test and control groups will fill out questionnaires before and after training to see changes in confidence and coping skills before and after training.

ELIGIBILITY:
Inclusion Criteria:

* the medical interns who participate in the education program for medical interns, who will work as interns at Seoul National University Hospital from March 2024
* participants who agree to the purpose of the study and consent to participation

Exclusion Criteria:

* who do not consent to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-04-13 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
self-rated confidence for managing emergency situation | 1 hour after education program
  self-rated confidence survey (10-Likert scale) for managing emergency situation: "I am confident in managing desaturation patients" 1: strongly disagree, 10: strongly agree
self-rated confidence for managing emergency situation | 6 months after starting intern training
  self-rated confidence survey (10-Likert scale) for managing emergency situation: "I am confident in managing desaturation patients" 1: strongly disagree, 10: strongly agree
performance in managing emergency situation | 1 week after education program
  Objective Structured Clinical Examination for physician's performance in managing emergency situation

SECONDARY OUTCOMES:
usability of Virtual Reality simulation program using User Experience Questionnaire Short | 1hour after education program
  usability survey of Virtual Reality simulation program using User Experience Questionnaire Short (7-Likert Scale: 1= negative, 7= positive)
usability of Virtual Reality simulation program using Simulator Sickness Questionnaire | 1hour after education program
  usability survey of Virtual Reality simulation program using Simulator Sickness Questionnaire (0:none, 1: slight, 2:moderate, 3:severe)
usability of Virtual Reality simulation program using System Usability Scale | 1hour after education program
  usability survey of Virtual Reality simulation program using System Usability Scale (5-Likert Scale: 1=strongly disagree, 5=strongly agree)